CLINICAL TRIAL: NCT05868018
Title: Evidence-based Practice Confidence and Behavior Throughout the Curriculum of Four Physical Therapy Education Programs: A Longitudinal Study
Brief Title: EBP Confidence and Behavior Throughout PT Edu
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Sacred Heart University (Other); University of Toronto (Other); Chatham University (Other)
Responsible Party: Principal Investigator, Judith E Deutsch, PT, PhD, Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro20140000413
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Evidence Based Practice; Physical Therapy; Education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DPT A: Students from University A received their typical evidence based practice education over 3 years.
  Interventions: Behavioral: Education
- DPT B: Students from University B received their typical evidence based practice education over 3 years.
  Interventions: Behavioral: Education
- DPT C: Students from University C received their typical evidence based practice education over 3 years.
  Interventions: Behavioral: Education
- MSPT: Students from University D received their typical evidence based practice education over 2 years.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — This was an observational study of changes in evidence based confidence and behavior across 4 physical therapy programs. Students received their typical physical therapy education and we measured changes in evidence based practice confidence and behaviors across programs throughout the curriculum.

SUMMARY:
This study aimed to describe changes in EBP confidence and behavior of students from four physical therapy education programs throughout their curriculum using the Evidence-Based Practice Confidence (EPIC) Scale and the Evidence-Based Practice Implementation Scale (EBPIS).

DETAILED DESCRIPTION:
Introduction Evidence-based practice (EBP) is a foundational process taught in health professional education, yet it is unclear when EBP confidence and skills are obtained.

Review of Literature Increases in EBP confidence and behaviors from the start of physical therapy programs to post graduation have been reported in studies that evaluated a single program or used non-valid questionnaires. This study aimed to describe changes in EBP confidence and behavior of students from four physical therapy education programs throughout their curriculum.

Subjects Two hundred sixty-nine physical therapy students were recruited across 4 PT programs (3 in US and 1 in Canada).

Methods Students completed the Evidence-Based Practice Confidence (EPIC) Scale and the Evidence-Based Practice Implementation Scale (EBPIS) at 6 timepoints: start of the program, prior to first clinical experience, after first clinical experience, at the end of classroom instruction, graduation, and one year post. Medians (Mdn) and 25th and 75th percentiles (P25, P75) were calculated for 42 (23.2%) students with complete data across all timepoints. Change between timepoints was assessed using Friedman's test and Wilcoxon signed rank test with a Bonferroni correction for post hoc analysis.

ELIGIBILITY:
Inclusion Criteria:

* students enrolled in the 4 selected physical therapy programs

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be enrolled in masters (University of Toronto) or doctorate physical therapy programs (Rutgers, Sacred Heart and Chatham). Physical therapy students and recent graduates will be invited to participate. Ages for students may range from 21-65
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Evidence Based Practice Confidence | 4 years
  10 item questionnaire
Evidence Based Practice Behavior | 3 years
  18 item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Romney, PhD, Study Director — Sacred Heart University

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified and shared with the study team.